CLINICAL TRIAL: NCT00839033
Title: Evaluation of a Mechanical Insufflation-exsufflation Device During Acute Respiratory Failure in Patients With Neuromuscular Disorders: a Prospective, Randomized, Controlled, Multicenter Study
Brief Title: Evaluation of a Mechanical Device During Acute Respiratory Failure in Patients With Neuromuscular Disorders
Acronym: Nemucough
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: No inclusion
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P080406
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Duchenne Muscular Dystrophy; Amyotrophic Lateral Sclerosis; Neuromuscular Diseases
Keywords: Cough assisted device; Neuromuscular disease; Respiratory exacerbation; Invasive ventilation,; Chest physiotherapy; Congenital myopathies
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Amyotrophic Lateral Sclerosis; Neuromuscular Diseases; Myotonia Congenita

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): patients treated with standard treatment and a mechanical insufflation-exsufflation
  Interventions: Device: mechanical insufflation - exsufflation
- 2 (Active Comparator): Patients with standard treatment and standard respiratory physiotherapy
  Interventions: Device: Standard respiratory physiotherapy

INTERVENTIONS:
Device: mechanical insufflation - exsufflation — Patients will receive MI-E treatment with the following settings: insufflation pressure of at least +30 cm H2O and an exsufflation pressure ≥ -30 cm H2O. There will be at least 6 hyperinflation/exsufflation sequences per session of chest physiotherapy. There will be at least two daily sessions done routinely by the respiratory therapist at 8 hour intervals.
  Other Names: Mechanical insufflation-exsufflation devices assist cough
  Arms: 1
Device: Standard respiratory physiotherapy — Traditional chest physiotherapy without mechanical insufflation-exsufflation
  Arms: 2

SUMMARY:
The hypothesis is that a mechanical insufflation-exsufflation (MI-E) is associated with a decrease in the number of intubations and more rapid clinical improvement in children and adults with neuromuscular disease who are admitted for an acute respiratory exacerbation.In this prospective, randomised, multicenter study, 55 patients will be treated with standard treatment and a MI-E, and 55 patients with standard treatment and standard respiratory physiotherapy. The primary objective is the reduction of the number of patients requiring invasive ventilatory support (endotracheal intubation or tracheotomy) in the group treated with MI-E (MI-E group). The main secondary objectives are a reduction in hospital stay and an improvement in clinical condition, dyspnea and respiratory muscle function.

DETAILED DESCRIPTION:
Justification Respiratory muscle weakness reduces the efficacy of the cough reflex in patients with neuromuscular disorders and exposes them to the risk of acute respiratory failure. Mechanical insufflation-exsufflation devices assist cough and have been shown to be efficient in increasing the cough expiratory flow in children and adults with neuromuscular disease and decreasing the risk of intubation in a limited population of hospitalized adults with acute respiratory failure.

Primary objective The goal is to record the efficacy of mechanical insufflation-exsufflation (MI-E) during acute respiratory failure in patients with neuromuscular disorders.The primary objective is the reduction of the number of patients requiring invasive ventilatory support (endotracheal intubation or tracheotomy) in the group treated with MI-E (MI-E group) compared to the group treated with traditional chest physiotherapy without MI-E (Control group).

Secondary objectives

In the MI-E group, compared to the Control group:

1. Decrease in the length of hospitalization in the intensive care unit (ICU)
2. Decrease in the total length of hospitalization
3. Decrease in the incidence of bronchoscopy-assisted aspiration
4. Decrease in the duration of oxygen therapy
5. Decrease in the daily length of noninvasive positive pressure ventilation (NPPV)
6. Improvement in blood gases on room air during hospitalization
7. Improvement of the peak cough flow (PCF)
8. Improvement of the vital capacity (VC), maximal inspiratory (PImax) and expiratory (PEmax) pressures, sniff nasal inspiratory pressure (SNIP), peak expiratory flow (PEF) and dyspnea during hospitalization.
9. Decrease in the number of secondary tracheotomies (for weaning of ventilatory support)

Type of study Prospective, randomized, controlled, multicenter study

Number of subjects The calculation of the number of subjects is based on two retrospective studies. In the study by VIANELLO, which included 11 adults hospitalized in the ICU for respiratory failure, the number of therapeutic failures, defined as the need for a "mini" tracheotomy or intubation, was significantly less in the group using MI-E than in a group of 16 historical control patients [2 failures in the MI-E group (18%) versus 10 failures in the control group (63%), p<0.05] (1). Another study reported 19 successes (80%) versus 5 failures on MI-E (2).

ELIGIBILITY:
Inclusion Criteria:

Pediatric or adult patients with chronic neuromuscular disorders, such as spinal muscular atrophy, Duchenne muscular dystrophy, other congenital myopathy, or amyotrophic lateral sclerosis (ALS), hospitalized for acute respiratory failure, as defined by:

* Persistent bronchial encumbrance (> 2 days) despite regular treatment in the homecare setting, associated with-Oxygen desaturation on room air, defined by a pulse oximetry (SaO2) <95%) or
* In patients not receiving long-term NPPV: the need to institute NPPV-In patients receiving long-term NPPV: the need to increase the daily length of NPPV by at least 25%.

Exclusion Criteria:

* Need for immediate intubation (alteration in consciousness, coma, hemodynamic disorders)
* Multiple organ failure (e.g., associated cardiac failure)
* In adults: respiratory rate >30/min, pH < 7.35, PaCO2 > 50 mm Hg
* Facial deformity or anomaly which prevents the use of a mouthpiece or mask
* Patients who signed a refusal to be intubated regardless of the progression of their disease
* Patients on long-term oxygen therapy
* Tracheotomized patients
* Patients requiring the use of an intrapulmonary percussive ventilation device during hospitalization
* Acute neuromuscular disorder of known or unknown etiology
* Associated lung disease such as chronic obstructive pulmonary disease (COPD)
* Refusal of patient consent and/or parental consent in the case of a minor
* Uncooperative patients
* Patients < 4 years old

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-06; Primary Completion 2011-02 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Reduction of the number of patients requiring invasive ventilatory support in the group treated with MI-E (MI-E group) compared to the group treated with traditional chest physiotherapy without MI-E (Control group). | During the treatment phase

SECONDARY OUTCOMES:
Decrease in the length of hospitalization in the intensive care unit (ICU) (if necessary) | During the treatment phase
Decrease in the total length of hospitalization | During the treatment phase
Decrease in the incidence of bronchoscopy-assisted aspiration | During the treatment phase
Decrease in the duration of oxygen therapy | During the treatment phase
Decrease in the daily length of noninvasive positive pressure ventilation (NPPV) | During the treatment phase
Improvement in blood gases on room air during hospitalization and improvement of the peak cough flow (PCF) | During the treatment phase
Improvement of the vital capacity (VC), maximal inspiratory (PImax) and expiratory (PEmax) pressures, sniff nasal inspiratory pressure (SNIP), peak expiratory flow (PEF) and dyspnea during hospitalization | During the treatment phase
Decrease in the number of secondary tracheotomies (for weaning of ventilatory support) | During the treatment phase

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte FAUROUX, MD PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hospital Armand Trousseau, Pediatric Pulmonology Department and INSERM UMR S-893, Paris, France